CLINICAL TRIAL: NCT01100918
Title: Utility of Tissue Doppler Echocardiography for Selecting Patients for Cardiac Resynchronisation Therapy in Heart Failure
Brief Title: Utility of Tissue Doppler Echocardiography for Selecting Patients for Cardiac Resynchronisation Therapy
Acronym: TIBI-HF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 004844BLT
Record Dates: First submitted 2010-04-08; First posted 2010-04-09 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Heart Failure
Keywords: Cardiac resynchronisation therapy; Tissue Doppler Imaging; Dyssynchrony
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1: Dyssynchrony positive (Active Comparator)
  Interventions: Device: BiV ICD
- 2a: Dyssynchrony negative (Active Comparator)
  Interventions: Device: BiV ICD
- 2b: Dyssynchrony negative (Active Comparator)
  Interventions: Device: ICD

INTERVENTIONS:
Device: BiV ICD — Biventricular ICD
  Arms: 1: Dyssynchrony positive; 2a: Dyssynchrony negative
Device: ICD — Implantable Defibrillator
  Arms: 2b: Dyssynchrony negative

SUMMARY:
Currently the main selection tool for Cardiac Resynchronisation Therapy (CRT) is the QRS duration on the surface echocardiography (ECG) which has been shown to be a poor predictor of response. We sought to evaluate the use of tissue Doppler (TDI) assessment of dyssynchrony in prediction of response to CRT.

The hypothesis is that the presence of mechanical dyssynchrony (measured using TDI echocardiography) successfully identifies heart failure patients who will respond to CRT. Conversely, the absence of mechanical dyssynchrony is associated with a low/no response to CRT.

This is a three arm study. Group 1 comprises patients with dyssynchrony on TDI who are implanted with a biventricular ICD whereas Group 2 patients comprise patients who have no dyssynchrony. Group 2 patients are randomised 1:1 to either receive a biventricular ICD (2a) or an ICD (2b). All patients undergo a NYHA class assessment, a cardiopulmonary exercise test, and an echocardiogram at baseline and at 6 months follow up. Baseline and 6 months findings will be compared in all three groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have an indication for ICD therapy
2. Heart failure of any aetiology with evidence of left ventricular (LV) systolic dysfunction with LV ejection fraction < 35% and LV cavity dilatation (end diastolic dimension > 55 mm)
3. NYHA Class III/IV symptoms of heart failure despite optimal medical therapy
4. QRS duration ≥120ms

Exclusion Criteria:

1. Reversible cause of heart failure such as ongoing ischaemia amenable to revascularisation or treatable valvular disease
2. Requirement for ventricular pacing due to atrioventricular block.
3. Limited life expectancy (< 6 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-02; Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary Exercise Testing - changes in Peak VO2 from baseline to 6 months | 6 months

SECONDARY OUTCOMES:
Change in New York Heart Association (NYHA) class from baseline to 6 months | 6 months
Change in Quality-of-Life score from baseline to 6 months | 6 months
Echocardiography - changes in left ventricular (LV) volume and dimensions, calculated ejection fractions and in severity of MR | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Schilling, MD, FRCP, Principal Investigator — Barts and the London NHS Trust, Queen Mary University of London
Locations (1):
- Barts and the London NHS Trust, London, United Kingdom